CLINICAL TRIAL: NCT03566095
Title: Voices for Food: Utilizing Food Policy Councils to Bridge the Gap Between Food Security and Healthy Food Choices
Brief Title: Voices for Food: Food Policy Councils, Food Security and Healthy Food Choices
Acronym: VFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Dakota State University (Other)
Collaborators: Michigan State University (Other); Ohio State University (Other); University of Nebraska Lincoln (Other); Purdue University (Other); University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-69004-20401
Record Dates: First submitted 2018-05-24; First posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Food Security; Nutritive Value
Keywords: Rural; Food Policy Councils; Food Pantry; Community Coaching
MeSH Terms: interventions — Voice

STUDY DESIGN:
Intervention Model Description: All data were collected from both treatment an comparison communities at the same time points.
Who Masked: Participant
Masking Description: Participants were not aware of their status as a treatment or comparison community.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching and Voices for Food Kit (Active Comparator): The treatment communities received community coaching from an Extension Professional or Educator in the use of the Voices for Food kit.
  Interventions: Behavioral: Coaching and Voices for Food Kit
- Voices for Food Kit (Sham Comparator): The comparison community received the Voices for Food kit.
  Interventions: Behavioral: Voices for Food Kit

INTERVENTIONS:
Behavioral: Coaching and Voices for Food Kit — Community Coaching and Voices for Food Kit
  Arms: Coaching and Voices for Food Kit
Behavioral: Voices for Food Kit — Voices for Food Kit
  Arms: Voices for Food Kit

SUMMARY:
This study evaluates the effectiveness of coaching and Voices for Food materials on establishing Food Policy Councils (FPCs) and using guided client choice in rural food pantries to improve food security and diet quality among food pantry clients, and to improve the food environment in rural, midwestern food pantries. Half of the communities received coaching and the Voices for Food kit, the other half only received the Voices for Food kit.

DETAILED DESCRIPTION:
Community coaching is a a strategy that helps community leaders plan for and overcome challenges to community development. Interventions at the community level are most effective when they are conceived and led by locals. Community coaches can aid the local community in the development of FPCs in rural communities. FPCs have the potential to improve the nutritional quality of available food, and connect a diverse network of food system stakeholders from the public, private and nonprofit sectors, which includes local food pantries. Food pantry users are food insecure and avoid hunger by consuming low cost and shelf stable food items. Guided client choice is a system of distribution that can be employed in food pantries and supported by FPCs. Guided client-choice is a model of distribution in which pantry clients choose the foods they would like from the pantry based upon family size and is formatted based upon USDA MyPlate. Guided client choice has been shown to meet the needs of the pantry client base better than the traditional model of distribution often found in food pantries. Food pantries have the opportunity to meet the nutritional needs of the food insecure population.

Voices for Food is a multi-leveled socio-ecological, longitudinal, matched treatment and comparison study to develop food policy councils (FPCs), and improve food security and diet quality in rural communities. Voices for Food was conducted in 24 rural, high poverty counties in South Dakota, Indiana, Missouri, Michigan, Nebraska and Ohio. Counties were assigned to a treatment (n=12) or comparison (n=12) group.

Intervention activities focus on three key components that impact food security: 1) community coaching by Extension Educators/field staff, 2) FPC development, and 3) development of a MyChoice (guided client choice) food pantry. Community coaching, along with the Voices for Food kit was only provided to treatment counties. Comparison communities only received the Voices for Food kit. Evaluation components focus on three levels of the intervention: 1) Community (FPCs), 2) Food Pantry Organization and Food Environment, and 3) Pantry Client & Families. Participants in this study were community stakeholders, food pantry directors, staff/volunteers and food pantry clients. Pantry food access/availability including pantry food quality and quantity, household food security and pantry client dietary intake are dependent variables.

ELIGIBILITY:
Inclusion Criteria:

* Food Pantry Clients must be current clientele by visiting the participating food pantry at least once in the last year, English-speaking.
* Food Pantry Directors must be 18 years or older (19 if in Nebraska), English-speaking and a director of a participating food pantry.
* Food Pantry Staff/Volunteers must be 18 years or older (19 if in Nebraska), English-speaking and a staff/volunteer of a participating food pantry.
* Community Stakeholders must be 18 years or older (19 if in Nebraska), English-speaking and reside in the participating community.

Exclusion Criteria:

* Under 18 years old (19 if in Nebraska)
* Non English- speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1735 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
The United States Household Food Security Survey Module | 4 years
  Change in food security of food pantry clients. Individuals will be classified as very low food secure, low food secure, marginal food secure and high food secure.
Healthy Eating Index (HEI) Score | 4 years
  Change in diet quality of food pantry clients. The Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Too allows for calculation of the Healthy Eating Index score, which is a measure of diet quality.

SECONDARY OUTCOMES:
Food Policy Council Implementation Form | 4 years
  The Food Policy Council Implementation Form is a study developed assessment tool that assesses the degree of food policy council implementation. The Food Council Implementation Form documents changes occurring within the Food Policy Council.
Food Pantry MyChoice Observation Tool | 4 years
  The Food Pantry MyChoice Observation Tool is a study developed assessment tool that assesses the degree of MyChoice (guided client choice) implementation. The tool documents the extent to which key components of the MyChoice food pantry model are physically in place at the pantry and part of the food, food display, and distribution process.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Stluka, PhD, RD, LN, Principal Investigator — South Dakota State University; Heather Eicher- Miller, PhD, Principal Investigator — Purdue University; Rebecca Henne, MS, Principal Investigator — Michigan State University; Donna Mehrle, MPH, RD, LD, Principal Investigator — University of Missouri-Columbia; Lisa Franzen-Castle, PhD, Principal Investigator — University of Nebraska Lincoln; Dan Remley, PhD, Principal Investigator — Ohio State University

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Wright BN, Vasquez-Mejia CM, Guenther PM, McCormack L, Stluka S, Franzen-Castle L, Henne B, Mehrle D, Remley D, Eicher-Miller HA. Fruit and Vegetable Healthy Eating Index Component Scores of Distributed Food Bags Were Positively Associated with Client Diet Scores in a Sample of Rural, Midwestern Food Pantries. J Acad Nutr Diet. 2021 Jan;121(1):74-83. doi: 10.1016/j.jand.2020.09.033. Epub 2020 Oct 21. PMID 33350943
- [Derived] Wright BN, Tooze JA, Bailey RL, Liu Y, Rivera RL, McCormack L, Stluka S, Franzen-Castle L, Henne B, Mehrle D, Remley D, Eicher-Miller HA. Dietary Quality and Usual Intake of Underconsumed Nutrients and Related Food Groups Differ by Food Security Status for Rural, Midwestern Food Pantry Clients. J Acad Nutr Diet. 2020 Sep;120(9):1457-1468. doi: 10.1016/j.jand.2020.04.011. Epub 2020 Jul 20. PMID 32703690
- [Derived] Liu Y, Tooze JA, Zhang Y, Leidy HJ, Bailey RL, Wright B, Ma M, Stluka S, Remley DT, McCormack LA, Franzen-Castle L, Henne R, Mehrle D, Eicher-Miller HA. Breakfast Consumption Is Positively Associated with Usual Nutrient Intakes among Food Pantry Clients Living in Rural Communities. J Nutr. 2020 Mar 1;150(3):546-553. doi: 10.1093/jn/nxz258. PMID 31711170
- [Derived] Stluka S, Moore L, Eicher-Miller HA, Franzen-Castle L, Henne B, Mehrle D, Remley D, McCormack L. Voices for food: methodologies for implementing a multi-state community-based intervention in rural, high poverty communities. BMC Public Health. 2018 Aug 23;18(1):1055. doi: 10.1186/s12889-018-5957-9. PMID 30139336